CLINICAL TRIAL: NCT02976883
Title: A Phase II, Single Centre Exploratory Study of [18F]HX4 PET/CT Imaging to Detect Hypoxia in Patients With Head and Neck and Lung Cancer, Receiving Radiotherapy With Curative Intent
Brief Title: [18F]HX4 PET/CT Imaging for Detection of Hypoxia
Acronym: OXYPET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13MP003
Record Dates: First submitted 2016-08-24; First posted 2016-11-29 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Head and Neck Cancer; Lung Cancer
Keywords: Hypoxia; HX4; PET CT; Radiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms; Lung Neoplasms; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [18F]HX4 diagnostic PET/CT scan (Experimental): [18F]HX4 (370 MBq) will be administered by a single intravenous injection, after which patients will be required to wait for ≤4.0 h and undergo a PET/CT scan.
  Interventions: Other: [18F]HX4 diagnostic PET/CT scan

INTERVENTIONS:
Other: [18F]HX4 diagnostic PET/CT scan — Single intravenous injection of [18F]HX4 and PET/CT scan

SUMMARY:
The aim of this study is to investigate the radiotracer [18F]HX4 for non-invasive detection of hypoxia in patients with head and neck, or lung cancer. Each participant will undergo a diagnostic [18F]HX4 PET/CT scan before beginning radiotherapy treatment. Patient follow up data will be collected from routine appointments, and analysed with the hypoxia scan results to assess whether [18F]HX4 PET/CT scanning can predict patient outcome from radiotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with:

  1. biopsy proven non-small cell carcinoma of the lung >2.5 cm in size with any T and N status but M0 who have elected to undergo radical radiotherapy or chemo-radiotherapy with curative intent or
  2. squamous cell carcinoma of the upper aerodigestive tract with a primary tumour or nodal mass >2. 5 cm in size, with any T and N status but M0 who have elected to undergo radical radiotherapy or chemo-radiotherapy with curative intent.
* Participant must be willing and able to give informed consent for participation in the study.
* Patients must be 18 years old or above.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
* Have normal renal function, defined by creatinine clearance of >60 mL/min.
* Able to remain still in the supine position on the scanner bed for the 40 minute duration of the examination.
* Able (in the Investigators opinion) and willing to comply with all study requirements.
* Willing to allow his or her General Practitioner and hospital consultant, if appropriate, to be notified of participation in the study

Exclusion criteria

* Patients who are scheduled for surgery prior to radiotherapy will not be included.
* Female participant who is pregnant, lactating or planning pregnancy during the course of the study.
* Chronic kidney disease stage III or worse, as defined by the NKF clinical practice guidelines (GFR <60 mL/min per 1.73 m3 for 3 months or more).
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of involvement in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Participants who have been involved in another research study involving an investigational product in the past 12 weeks.
* Previous surgery or radiotherapy to the upper aerodigestive tract or lung, which in the opinion of the Investigators could compromise the data.
* Previous cancer diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-03-31 (Actual); Primary Completion 2017-07-25 (Actual); Study Completion 2017-07-25 (Actual)

PRIMARY OUTCOMES:
The number of participants with primary treatment failure, tumour recurrence, disease free survival in the first two years after radiotherapy | 2 years

SECONDARY OUTCOMES:
Collection of outcome data to determine number of participants with tumour recurrence or disease free survival 5 years after radiotherapy treatment. | 5 years
Comparison of measurements of tumour/nodal disease areas on pre-treatment [18F]FDG PET/CT images with [18F]HX4 PET/CT images | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Alan C Perkins, PhD, Study Chair — Nottingham University Hospitals NHS Trust
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided